CLINICAL TRIAL: NCT06547437
Title: "Evaluating the Effectiveness of Papaverine as an Adjunct to Oxytocin for Labor Induction: A Randomized Controlled Trial"
Brief Title: Papaverine and Oxytocin vs Oxytocin Alone in Labor Induction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Inshirah Sgayer, DR inshirah sgayer galilee medical center, Western Galilee Hospital-Nahariya
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0124-24-NHR
Record Dates: First submitted 2024-08-01; First posted 2024-08-09 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Induced; Birth; Labor Onset and Length Abnormalities
MeSH Terms: interventions — Papaverine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Intervention Group: Combined use of papaverine (80 mg intravenous mg in 100 mL saline once concurrent with the start of oxytocin) and oxytocin.
  Control Group: Oxytocin plus 100 mL saline.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blinded study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- oxytocin plus papaverine (Active Comparator): Intervention Group: Combined use of papaverine (80 mg intravenous mg in 100 mL saline once concurrent with the start of oxytocin) and oxytocin.
  Interventions: Drug: Papaverine
- oxytocin alone (Placebo Comparator): Control Group: Oxytocin plus 100 mL saline.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Papaverine — papaverine a smooth muscle relaxant
  Arms: oxytocin plus papaverine
Drug: normal saline — normal saline 0.9% 100 cc
  Other Names: normal saline 0.9% 100 cc
  Arms: oxytocin alone

SUMMARY:
This study aims to evaluate the efficacy and safety of combining papaverine with oxytocin for labor induction compared to oxytocin alone

DETAILED DESCRIPTION:
Labor induction is a common obstetric procedure aimed at stimulating uterine contractions to initiate labor, often due to medical or obstetric indications such as post-term pregnancy, preeclampsia, or fetal growth restriction. The primary objective is to achieve vaginal delivery while minimizing risks to both mother and child. Oxytocin, a synthetic analog of the natural hormone, is the most frequently used pharmacological agent for labor induction due to its effectiveness in promoting uterine contractions. However, its use is associated with complications, including uterine hyperstimulation, increased need for epidural analgesia, and higher rates of operative deliveries.

The potential of antispasmodics to aid in labor induction has been explored, with some studies indicating that these agents can reduce the duration of labor and enhance cervical dilation. The Cochrane review on antispasmodics for labor highlighted that these drugs, such as hyoscine butylbromide and drotaverine, could significantly reduce the duration of the first stage of labor and increase the rate of cervical dilation, although the overall quality of evidence was low. Despite these findings, further high-quality studies are recommended to substantiate these benefits and ensure safety.

Papaverine, a well-known smooth muscle relaxant traditionally used for treating vascular spasms, presents a promising adjunctive therapy for labor induction. By relaxing the smooth muscles of the cervix and uterus, papaverine may facilitate more efficient cervical ripening and enhance the effectiveness of oxytocin-induced contractions. Preliminary studies with other antispasmodics, such as butylscopolamine, have shown reductions in labor duration and improvements in labor progression without significant adverse effects, suggesting that papaverine might offer similar benefits.

This study aims to evaluate the efficacy and safety of combining papaverine with oxytocin for labor induction compared to oxytocin alone. The primary outcome will be the time to onset of active labor, with secondary outcomes including total duration of labor, rate of cesarean deliveries, maternal satisfaction, and adverse effects. By investigating this novel combination, the study seeks to provide new insights into optimizing labor induction protocols, ultimately improving maternal and neonatal outcomes.

Objective: To evaluate if adding papaverine to oxytocin reduces the time to active labor compared to oxytocin alone.

Design: a randomized controlled study Participants: Pregnant women at term requiring labor induction using oxytocin. Intervention Group: Combined use of papaverine (80 mg intravenous mg in 100 mL saline once concurrent with the start of oxytocin) and oxytocin.

Control Group: Oxytocin plus 100 mL saline.

Primary outcome: Time to onset of active labor. Secondary outcomes: Total duration of labor, length of first stage of labor, length of second stage of labor, rate of cesarean deliveries, rate of cervical dilation.

ELIGIBILITY:
Inclusion Criteria:

* Women with a singleton pregnancy Over the age of 18 Term (between 37-42 weeks of gestation) A medical decision for labor induction using oxytocin. Cephalic presentation Viable fetus nulliparity

Exclusion Criteria:

* parity >1
* Twin pregnancy Women with a previous cesarean section Severe fetal anomalies Women with psychiatric disorders, including depression and schizophrenia. Contraindication to vaginal delivery Women unable to sign the consent form Women known to have SVT (supraventricular tachycardia). Women with a heart rate over 100 or arrhythmia Known sensitivity to any component of the drug Liver disease

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 126 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
time to active delivery | 24 HOURS AFTER DELIVERY
  time from labor induction till dilatation of 6 cm

SECONDARY OUTCOMES:
vaginal deliveries in 24 hours | 24 HOURS AFTER DELIVERY
  rate of vaginal deliveries in 24 hours
total length of labor | 24 HOURS AFTER DELIVERY
  time for induction to delivery
cesarean delivery rate | ho24 HOURS AFTER DELIVERY
  rate of emergent cesarean delivery during labor
length of second stage of labor | 24 hours after delivery
  second stage of labor in hours

IPD SHARING:
Plan to Share IPD: Undecided